CLINICAL TRIAL: NCT04017962
Title: An Open-label, Single-arm Study of Letermovir (LTV) for Prevention of Recurrent CMV Infection in High-risk Hematopoietic Cell Transplant (HCT) Recipients
Brief Title: A Study of the Drug Letermovir (LTV) as Prevention for Recurrent of Cytomegalovirus (CMV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-174
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: CMV; CMV Infection; Hematopoietic Cell Transplant
Keywords: HCT; CMV infection; Letermovir; LTV; Memorial Sloan Kettering Cancer Center; 19-174
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hematopoietic cell transplantation/HCT (Experimental): Participants will be hematopoietic cell transplantation (HCT) recipients with a history of CMV infection. INTERVENTIONAL COHORT: Patients receive letermovir PO QD (or IV over 1 hour for patients unable to receive PO) for 14 weeks in the absence of disease progression or unacceptable toxicity.
  OBSERVATIONAL COHORT: Patients undergo collection of blood samples for CMV-CMI analysis via CMV immunity T cell panel assay on day 100. Patients with negative CMI on day 100 undergo collection of blood samples for retesting on day 180.
  Interventions: Drug: Letermovir Pill; Other: blood draw

INTERVENTIONS:
Drug: Letermovir Pill — Patients enrolled on the study will receive oral LTV 480 mg daily (240 mg daily for patients receiving cyclosporine A). The maximum duration of LTV administration will be 14 weeks. Patients receiving oral medication will be administered a pill diary for drug compliance purposes. This will be administered and reconciled in clinic.
  Other Names: LTV
Other: blood draw — Collection of blood samples for CMV-CMI analysis via CMV immunity T cell panel assay on day 100. Patients with negative CMI on day 100 undergo collection of blood samples for retesting on day 180.

SUMMARY:
The purpose of this study is to determine of letermovir (LTC) is effective at preventing Cytomegalovirus (CMV) infection from returning in people who have already had CMV infection after a bone marrow transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 12 years (any weight)
* Have received allogenic HCT
* Have received preemptive therapy for clinically significant CMV infection post-HCT and have completed preemptive therapy no longer than 7 days prior to enrollment. Preemptive treatment includes ganciclovir, valganciclovir, foscarnet or cidofovir. Clinically significant CMV infection is defined as CMV viremia requiring preemptive therapy or CMV EOD. Patients who have received LTV prophylaxis prior to onset of clinically significant CMV infection prior to enrollment (see also exclusion criteria below).
* Have one or more risk factors for recurrent CMV infection:

  1. Human leukocyte antigen (HLA) mismatch

     * HLA-related (sibling) donor with at least one mismatch at the HLA-A, -B or -DR gene loci
     * Haploidentical donor
     * Unrelated donor with at least one mismatch at the HLA-A, -B, -C or -DRC1gene loci, or
     * Cord blood as stem cell source
  2. Acute or chronic GVHD requiring either topical steroids for gastrointestinal GVHD and/or systemic steroid treatment (>/= 1mg/kg/day of prednisone or equivalent dose of another corticosteroid) within 14 days prior to enrollment
  3. T-cell-depleted allograft ex-vivo or in-vivo T-cell depleting agents including but not limited to ATG, alemtuzimab and post HCT cyclophosphamide.
* For adult patients, able to provide written consent and complete the informed consent. For patients under 18 years, the patient's parent(s) or legal guardian(s) must provide informed consent and the patient must provide written assent to participation in the study.
* Willing and able to comply with trial instructions and requirements
* Male and female patients of childbearing potential must be willing to use a highly effective method of contraception for the course of the study. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Subject eligibility criteria for the observational cohort:

* Age 18 years or older
* First allogenic peripheral blood or marrow HCT
* LTV prophylaxis starting <30 days post HCT and given for at least 6 weeks

Exclusion Criteria:

* Clinically significant CMV infection present at enrollment
* Breakthrough CMV infection while on primary LTV prophylaxis (unless patient non-adherent or unable to adequately absorb letermovir or documented resistance to LTV.
* Glomerular filtration rate (GFR) </= mL/min/1.73m^2(equivalent to creatinine clearance </=10 mL/min)
* Severe hepatic impairment
* Routine use of high-dose acyclovir (doses of > 800 mg twice daily), valacyclovir (doses of > 500mg twice daily), or famciclovir (doses > 500mg/day) for varicella zoster virus (VZV)/herpes simplex virus prophylaxis; limited treatment courses at higher doses for VZV infections are permissible if treatment duration dose not exceed 14 days total. Short courses of IV cidofovir for adeno virus (ADV) are permissible
* Suspected or known hypersensitivity to active or inactive ingredients of LTV formulations
* Patients treated with a medication whose administration with LTV is ontraindicated and whose discontinuation is not possible. Contraindicated medications include pimozide, ergot alkaloids and pitavastatin or simvastatin when co-administered with cyclosporine.
* Imminent demise (expected survival <6 weeks)
* Documented positive result for human immunodeficiency virus antibody (HIV-Ab) or for hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) at any time prior to HCT
* Need for mechanical ventilation and/or vasopressor support at the time of enrollment
* Pregnancy or breastfeeding
* Plans to conceive or father children within the projected duration of the trial
* History of current evidence of any condition, therapy, lab abnormality, or other circumstance that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or would place the subject at undue risk as judged by the investigator, such that it is not in the best interest of the subject to participate in this study.
* The following antivirals are allowed up to the listed dose limits:

  * Acyclovir up to 800 mg twice daily
  * Valacyclovir up to 500 mg twice daily
  * Famciclovir up to 500 mg/day for VZV/HSV prophylaxis; limited treatment courses at higher doses for VZV infections are permissible if treatment duration does not exceed 14 days total.
  * Short courses of IV cidofovir for ADV (up to two doses)

Exclusion criteria for observational cohort:

* Clinically significant CMV infection during the 100 days following HCT. Clinically significant CMV infection defined as either CMV viremia requiring preemptive therapy with CMV antivirals or CMV end organ disease (EOD)
* Grade 3-4 GVHD
* Cord blood as cell source for HCT
* Treatment with systemic steroids (>0.5mg/kg for 2 weeks or longer) within 3 weeks prior to enrollment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2025-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genovefa Papanicolaou, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Related Info — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Cell Transplantation/HCT: INTERVENTIONAL COHORT: Patients receive letermovir PO QD (or IV over 1 hour for patients unable to receive PO) for 14 weeks in the absence of disease progression or unacceptable toxicity. Participants will be hematopoietic cell transplantation (HCT) recipients with a history of CMV infection.
- Observational Cohort: Participants will be hematopoietic cell transplantation (HCT) recipients with a history of CMV infection. Patients undergo collection of blood samples for CMV-CMI analysis via CMV immunity T cell panel assay on day 100. Patients with negative CMI on day 100 undergo collection of blood samples for retesting on day 180.
Period: Overall Study
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Started | 36 | 66
Completed | 26 | 66
Not Completed | 10 | 0
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Discontinued LTV | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort | Total
Number analyzed (Participants) | 36 | 66 | 102
Age, Continuous [Median (Full Range); unit: years] | 59 [17 to 84] | 63 [22 to 77] | 60 [17 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 18 | 37 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 10 | 14
  Not Hispanic or Latino | 32 | 56 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 22 | 50 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 66 | 101
  India | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant CMV Viremia for Hematopoietic Cell Transplantation/HCT Participants in the Interventional Cohort Only
Description: Clinically significant CMV viremia defined as: Any level CMV DNAemia requiring preemptive treatment per Institutional standard of care at each participating Institution.
Time Frame: 14 weeks
Population: Outcome measure relevant for Hematopoietic Cell Transplantation/HCT cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Number analyzed (Participants) | 36 | 0
Participants
  Participants with clinically significant CMV viremia | 5 | 0
  Participants without clinically significant CMV viremia | 31 | 0

2. Secondary Outcome: Number of Participants With Breakthrough Clinically Significant CMV Viremia With Emergence of Letermovir-resistant CMV Virus for Hematopoietic Cell Transplantation/HCT Participants in the Interventional Cohort Only
Description: Emergence of Letermovir-resistant CMV Virus in Patients with breakthrough clinically significant CMV viremia.
Time Frame: 14 weeks
Population: Outcome measure relevant for Hematopoietic Cell Transplantation/HCT cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Number analyzed (Participants) | 36 | 0
Participants
  Pts with breakthrough clinically significant CMV viremia and Letermovir-resistant CMV Virus | 2 | 0
  Pts w/breakthrough clinically significant CMV viremia w/out Letermovir-resistant CMV Virus | 2 | 0
  Pts without breakthrough clinically significant CMV viremia | 32 | 0

3. Secondary Outcome: CMV End Organ Disease for Hematopoietic Cell Transplantation/HCT Participants in the Interventional Cohort Only
Time Frame: 14 weeks
Population: Outcome measure relevant for Hematopoietic Cell Transplantation/HCT cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Number analyzed (Participants) | 36 | 0
Participants
  Pts with CMV end organ disease | 0 | 0
  Pts without CMV end organ disease | 36 | 0

4. Secondary Outcome: CMV Related Death for Hematopoietic Cell Transplantation/HCT Participants in the Interventional Cohort Only
Time Frame: 14 weeks
Population: Outcome measure relevant for Hematopoietic Cell Transplantation/HCT cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Number analyzed (Participants) | 36 | 0
Participants
  Pts with CMV related death | 0 | 0
  Pts without CMV related death | 36 | 0

5. Secondary Outcome: Adverse Events at Least Possibly Related to Letermovir by the Treating Physician for Hematopoietic Cell Transplantation/HCT Participants in the Interventional Cohort Only
Time Frame: 14 weeks
Population: Outcome measure relevant for Hematopoietic Cell Transplantation/HCT cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
Number analyzed (Participants) | 36 | 0
Participants
  Pts with AE's at least possibly related to Letermovir | 0 | 0
  Pts without AE's at least possibly related to Letermovir | 36 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Hematopoietic Cell Transplantation/HCT | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 2/36 | 0/66
Serious Adverse Events (participants affected / at risk) | 2/36 | 0/66
Other Adverse Events (participants affected / at risk) | 0/36 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hematopoietic Cell Transplantation/HCT (N=36) | Observational Cohort (N=66)
Death NOS (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04017962/Prot_SAP_000.pdf